CLINICAL TRIAL: NCT06966635
Title: Exploratory Study on the Treatment of Gout With Potassium Citrate Sustained-release Tablets
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhu Xiaoxia, Associate Chief Physician, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-641
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hyperuricemia or Gout; Nephrolithiasis
MeSH Terms: conditions — Hyperuricemia; Gout; Nephrolithiasis | interventions — Sodium Bicarbonate; Potassium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controll group (Active Comparator): The control group was treated with the standard uric acid-lowering treatment regimen alone. Uric acid-lowering treatment plan: Maintain the individualized uric acid-lowering treatment plan at the time of patient enrollment. Traditional uric acid-lowering treatment plans include drugs that reduce uric acid production such as febuxostat and allopurinol, and drugs that increase uric acid excretion such as benzbromarone.
  Interventions: Drug: uric-acid-lowering drug
- Potassium citrate group (Experimental): On the basis of the standard uric acid-lowering treatment plan, potassium citrate was taken three times a day, 2.16g each time.
  Interventions: Drug: Potassium Citrate Tablets; Drug: uric-acid-lowering drug
- Sodium bicarbonate group (Experimental): Sodium Bicarbonate Oral Capsule
  Interventions: Drug: Sodium Bicarbonate Oral Capsule; Drug: uric-acid-lowering drug

INTERVENTIONS:
Drug: Sodium Bicarbonate Oral Capsule — On the basis of the standard uric acid-lowering treatment plan, sodium bicarbonate should be taken three times a day, 1.0g each time
  Arms: Sodium bicarbonate group
Drug: Potassium Citrate Tablets — On the basis of the standard uric acid-lowering treatment plan, potassium citrate was taken three times a day, 2.16g each time
  Arms: Potassium citrate group
Drug: uric-acid-lowering drug — The control group was treated with the standard uric acid-lowering treatment regimen alone. Uric acid-lowering treatment plan: Maintain the individualized uric acid-lowering treatment plan at the time of patient enrollment. Traditional uric acid-lowering treatment plans include drugs that reduce uric acid production such as febuxostat and allopurinol, and drugs that increase uric acid excretion such as benzbromarone. At the time of enrollment, the uric acid-lowering drugs were stable. The treatment plan for lowering uric acid remained unchanged for 4 weeks after enrollment in the clinical study until the endpoint.

SUMMARY:
To evaluate whether alkalization has the effect of lowering uric acid and reducing gout flare and determine whether alkalization has a role in the prevention and treatment of urinary calculi in gout, the research participants were divided into the control group, the potassium citrate group and the sodium bicarbonate group. 2 alkalization groups took potassium citrate three times a day 2.16g each time, or sodium bicarbonate three times a day, 1.0g each time, on the basis of the standard uric acid-lowering treatment plan. The control group was treated with the standard uric acid-lowering treatment regimen alone. Uric acid-lowering treatment plan: Maintain the individualized uric acid-lowering treatment plan at the time of patient enrollment. Traditional uric acid-lowering treatment plans include drugs that reduce uric acid production such as febuxostat and allopurinol, and drugs that increase uric acid excretion such as benzbromarone. At the time of enrollment, the uric acid-lowering drugs were stable.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of the American College of Rheumatology (ACR) and the European League against Rheumatism (EULAR) for gout in 2015
* Age 18-70 years old, gender is not limited
* The interval between the most recent acute onset of gout is at least > 2 weeks
* Routine treatment with stable dose of uric-lowering drugs for > 4 weeks
* For women who are likely to become pregnant, pregnancy tests must be negative, they must not be lactating, they must be using an investigator-approved method of contraception, and they must agree to maintain this method of contraception throughout the study
* Study participants were informed, voluntarily signed informed consent, and agreed to participate in all visits, examinations, and treatments as required by the trial protocol
* Informed consent to the purpose and content of the research.

Exclusion Criteria:

* Acute gout flare
* Secondary gout caused by kidney disease, blood disease, or taking certain drugs, tumor radiotherapy and chemotherapy
* Severe and unstable cardiovascular and cerebrovascular diseases (such as unstable angina pectoris, coronary angiogenesis, cerebral angiogenesis, transient ischemic attack, congestive heart failure, etc.), acute and difficult to control diseases, chronic diffuse connective tissue disease, xanthine urethral deposition, Lesch-Nyhan syndrome, untreated thyroid disease or kidney stones, treatment Patients with severe hypertension (blood pressure > 160/100mmHg) or diabetes (fasting blood glucose > 11.1mmol/L) and organ transplantation that were not effectively controlled later
* People who are allergic, have a history of allergy to test-related drugs (febuxosita tablets, allopurinol tablets, benzbromarone, etoracoxib, colchicine, potassium citrate, etc.) or are allergic to test-related drug components
* Active peptic ulcer or ulcer with bleeding and perforation, severe chronic diarrhea or recurrent skin disease in the past year
* Blood white blood cell count < 3.0x109/L, hemoglobin < 90g/L, platelet count < 100x109/L, or other blood system diseases (such as severe anemia, idiopathic thrombocytopenic purpura, spleen enlargement, coagulation dysfunction, etc.)
* Active stage of liver disease or abnormal liver function (ALT or AST≥2 times the upper limit of normal)
* Patients with abnormal renal function (eGFR≤60ml/min/1.73m^2)
* Patients with elevated blood potassium (5.5mmol/L) may have diseases or factors that may lead to hyperkalemia, such as type IV renal tubular acidosis and widespread tissue injury
* Urine PH value > 6.5 during screening
* Combined use of the following drugs: Contains salicylate drugs such as aspirin (> 300mg/d), thiazide diuretics, potassium diuretics such as amphenopterine, Amiloride, ACEI, azathioprine, 6-mercaptopurine, theophylline, losartan, cyclosporin A, cyclophospfamide, pyrazinamide, glucocorticoid (except in acute episodes), Niergoline tablets, long-term use of insulin, Digitalis
* Women who are pregnant, planning to become pregnant or breastfeeding mental illness, no self-knowledge, unable to accurately express or can not take drugs on time
* A history of alcohol abuse or dependence on known drugs within the last two years
* Those who have participated or are participating in other clinical trials within three months
* The study participant is a family member or relative of the staff of the research Center
* Other lesions or conditions that, in the investigator's judgment, reduce or complicate enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
serum uric acid | From enrollment to the end of treatment at 48 weeks

SECONDARY OUTCOMES:
gout flare | From enrollment to the end of treatment at 48 weeks

OTHER OUTCOMES:
nephrolithiasis | From enrollment to the end of treatment at 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial. Contact the author by email after the research is completed.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results